CLINICAL TRIAL: NCT02734615
Title: A Phase I/Ib, Open Label Study of LSZ102 Single Agent and LSZ102 in Combination With Either LEE011 (LSZ102 + LEE011) or BYL719 (LSZ102 + BYL719) in Patients With Advanced or Metastatic ER+ Breast Cancer Who Have Progressed After Endocrine Therapy
Brief Title: Phase I/Ib Trial of LSZ102 Single Agent or LSZ102 + LEE011 or LSZ102 + BYL719 in ER+ Breast Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLSZ102X2101; 2015-004016-38 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Advanced or Metastatic ER+ Breast Cancer
Keywords: LSZ102; LEE011; ribociclib; Kisqali; BYL719; alpelisib; ER+ breast cancer; advanced ER+ breast cancer; metastatic ER+ breast cancer; SERD; SERM; fulvestrant; tamoxifen; aromatase inhibitor; ESR1; mtESR1; wtESR1; estrogen receptor; endocrine therapy
MeSH Terms: interventions — LSZ102; ribociclib; Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A (Experimental): Patients will get LSZ102 single agent during dose escalation.
  Interventions: Drug: LSZ102
- Arm B (Experimental): Patients will get LSZ102 in combination with LEE011 during dose escalation.
  Interventions: Drug: LSZ102; Drug: LEE011
- Arm C (Experimental): Patients will get LSZ102 in combination with BYL719 during dose escalation.
  Interventions: Drug: LSZ102; Drug: BYL719
- Arm 1 (Experimental): Patients will get LSZ102 single agent during dose expansion
  Interventions: Drug: LSZ102
- Arm 2 (Experimental): Patients will get LSZ102 + LEE011 (LEE011 intermittent regimen) during dose expansion
  Interventions: Drug: LSZ102; Drug: LEE011
- Arm 3 (Experimental): Patients will get LSZ102 + LEE011 (LEE011 continuous regimen) during dose expansion
  Interventions: Drug: LSZ102; Drug: LEE011
- Arm 4 (Experimental): Patient will get LSZ102 in combination with BYL719 during dose expansion
  Interventions: Drug: LSZ102; Drug: BYL719

INTERVENTIONS:
Drug: LSZ102 — LSZ102
Drug: LEE011 — LEE011
  Other Names: ribociclib, Kisqali
  Arms: Arm 2; Arm 3; Arm B
Drug: BYL719 — BYL719
  Other Names: alpelisib
  Arms: Arm 4; Arm C

SUMMARY:
To characterize the safety and tolerability, identify recommended doses and regimens for future studies, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of LSZ102 as a single agent and in combination with either LEE011 or BYL719 in adult patients with locally advanced or metastatic ER+ breast cancer who have progressed after endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any procedures
* Histologically and/or cytologically confirmed diagnosis of ER+/HER2- breast cancer
* Advanced or metastatic breast cancer
* Must be able to swallow tablets and capsules

Exclusion Criteria:

* Symptomatic CNS metastases
* Patients whose laboratory values do not meet protocol criteria
* Clinically significant cardiac disease
* Impaired gastrointestinal function (GI) or GI disease that may significantly alter the absorption of oral medications

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Day 1 - Day 28 of Cycle 1 (28 day cycle)
  The dose escalation part of the study will be guided by well-established statistical methods/models to estimate the maximum tolerated doses (MTD)and/or recommended doses for expansion (RDE). Safety, pharmacokinetic and pharmacodynamics data will guide dose escalation decisions.
Safety and tolerability of LSZ102, LSZ102 + LEE011 and LSZ102 + BYL719 | Approximately 3 years
  Incidence and severity of adverse events, serious adverse events, clinical laboratory values, vital signs, ECGs, dose interruptions, dose reductions and dose intensity.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Approximately 3 years
  Assessment of preliminary anti-tumor activity of LSZ102, LSZ102 + LEE011 and LSZ102 + BYL719. ORR is defined as the proportion of patients with a best overall response of complete response or partial response.
Duration of Response (DOR) | 3 years
  Assessment of preliminary anti-tumor activity of LSZ102, LSZ102 + LEE011 and LSZ102 + BYL719
Progression Free Survival (PFS) | 3 years
  Assessment of preliminary anti-tumor activity of LSZ102, LSZ102 + LEE011 and LSZ102 + BYL719
Disease control rate (DCR) | 3 years
  Assessment of preliminary anti-tumor activity of LSZ102, LSZ102 + LEE011 and LSZ102 + BYL719
Plasma concentration of study medications | 1 cycle (28 day cycle)
  Plasma concentration versus time
Plasma concentration under fasted condition and fed condition | Up to 2 cycles (28 day cycle)
  Plasma concentration versus time under fasted and fed conditions
Levels of Pharmacodynamic marker Estrogen receptor (ER) | 3 years
  To assess pharmacodynamics effect
Levels of Pharmacodynamic marker Progesterone receptor (PgR) | 3 years
  To assess the pharmacodynamic effect
Levels of Pharmacodynamic marker pS6 | 3 years
  To assess the pharmacodynamic effect
Pharmacokinetics (PK) parameter AUC | 6 cycles (28 day cycle)
  AUC = Area under curve
PK parameter Cmax | 6 cycles (28 day cycle)
  Cmax = Maximum observed plasma concentration after drug administration
PK parameter Tmax | 6 cycles (28 day cycle)
  Tmax = Time to reach Cmax
PK parameter Cmin | 6 cycles (28 day cycle)
  Cmin = Minimum observed plasma concentration after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (3):
  - Massachusetts General Hospital Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center SC - LSZ102X2101, Houston, Texas
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Ulm, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jhaveri K, Juric D, Yap YS, Cresta S, Layman RM, Duhoux FP, Terret C, Takahashi S, Huober J, Kundamal N, Sheng Q, Balbin A, Ji Y, He W, Crystal A, De Vita S, Curigliano G. A Phase I Study of LSZ102, an Oral Selective Estrogen Receptor Degrader, with or without Ribociclib or Alpelisib, in Patients with Estrogen Receptor-Positive Breast Cancer. Clin Cancer Res. 2021 Nov 1;27(21):5760-5770. doi: 10.1158/1078-0432.CCR-21-1095. Epub 2021 Aug 25. PMID 34433648
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17965